CLINICAL TRIAL: NCT00591474
Title: The Influence of Probiotics on Vancomycin-Resistant Enterococcus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant lost to followup
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Robert Martindale, MD, PhD, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB3848
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: GI Colonization of Vancomycin-resistant Enterococcus
Keywords: VRE; Probiotics; colonization; gut health
MeSH Terms: interventions — Probiotics; Yogurt

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): VRE positive patients
  Interventions: Dietary Supplement: probiotics
- 2 (Placebo Comparator): VRE positive patients
  Interventions: Dietary Supplement: yogurt

INTERVENTIONS:
Dietary Supplement: probiotics — 100 gms of a yogurt drink containing probiotics will be given to pVRE positive patients for 4 weeks
  Arms: 1
Dietary Supplement: yogurt — 100 gms of pasteurized yogurt drinks with no live cultures will be given to VRE positive patients for 4 weeks
  Arms: 2

SUMMARY:
Drinking probiotics in a the form of a yogurt drink will restore normal gastrointestinal (GI) bacteria in patients whose colon are colonized with vancomycin-resistant enterococcus (VRE).

ELIGIBILITY:
Inclusion Criteria:

* VRE positive patients with GI colonization

Exclusion Criteria:

* Age less than 18 years
* Patients who have had a bone marrow transplant
* Extreme short bowel patients (less than 100 cm small bowel remaining)
* Patients with active VRE infection but no GI colonization
* Patients unable to eat and have no feeding access
* Patients who do not have a power of attorney to give consent if they are unable to

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Whether a positive VRE colonized patient becomes VRE negative after drinking yogurt with probiotics | 4 weeks

SECONDARY OUTCOMES:
Time to VRE clearance | 4 weeks
Sustainable effects of probiotics on VRE colonization | 8 weeks
Any positive or negative effects on patients' hospital stay. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martindale, MD, PH.D, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU hospital, Portland, Oregon, United States

REFERENCES:
- [Background] Zirakzadeh A, Patel R. Vancomycin-resistant enterococci: colonization, infection, detection, and treatment. Mayo Clin Proc. 2006 Apr;81(4):529-36. doi: 10.4065/81.4.529. PMID 16610573
- [Background] National Nosocomial Infections Surveillance System. National Nosocomial Infections Surveillance (NNIS) System Report, data summary from January 1992 through June 2004, issued October 2004. Am J Infect Control. 2004 Dec;32(8):470-85. doi: 10.1016/S0196655304005425. No abstract available. PMID 15573054
- [Background] Harbarth S, Cosgrove S, Carmeli Y. Effects of antibiotics on nosocomial epidemiology of vancomycin-resistant enterococci. Antimicrob Agents Chemother. 2002 Jun;46(6):1619-28. doi: 10.1128/AAC.46.6.1619-1628.2002. No abstract available. PMID 12019066
- [Background] Joels CS, Matthews BD, Sigmon LB, Hasan R, Lohr CE, Kercher KW, Norton J, Sing RF, Heniford BT. Clinical characteristics and outcomes of surgical patients with vancomycin-resistant enterococcal infections. Am Surg. 2003 Jun;69(6):514-9. PMID 12852510
- [Background] Pelz RK, Lipsett PA, Swoboda SM, Diener-West M, Powe NR, Brower RG, Perl TM, Hammond JM, Hendrix CW. Vancomycin-sensitive and vancomycin-resistant enterococcal infections in the ICU: attributable costs and outcomes. Intensive Care Med. 2002 Jun;28(6):692-7. doi: 10.1007/s00134-002-1276-8. Epub 2002 Apr 12. PMID 12107672
- [Background] Weinstock DM, Conlon M, Iovino C, Aubrey T, Gudiol C, Riedel E, Young JW, Kiehn TE, Zuccotti G. Colonization, bloodstream infection, and mortality caused by vancomycin-resistant enterococcus early after allogeneic hematopoietic stem cell transplant. Biol Blood Marrow Transplant. 2007 May;13(5):615-21. doi: 10.1016/j.bbmt.2007.01.078. Epub 2007 Mar 23. PMID 17448922
- [Background] Matar MJ, Tarrand J, Raad I, Rolston KV. Colonization and infection with vancomycin-resistant Enterococcus among patients with cancer. Am J Infect Control. 2006 Oct;34(8):534-6. doi: 10.1016/j.ajic.2006.04.205. PMID 17015161
- [Background] Humphreys H, Dolan V, Sexton T, Conlon P, Rajan L, Creamer E, Walshe J, Donohoe J, Smyth EG. Implications of colonization of vancomycin-resistant enterococci (VRE) in renal dialysis patients. Learning to live with it? J Hosp Infect. 2004 Sep;58(1):28-33. doi: 10.1016/j.jhin.2004.04.022. PMID 15350710
- [Background] Zaas AK, Song X, Tucker P, Perl TM. Risk factors for development of vancomycin-resistant enterococcal bloodstream infection in patients with cancer who are colonized with vancomycin-resistant enterococci. Clin Infect Dis. 2002 Nov 15;35(10):1139-46. doi: 10.1086/342904. Epub 2002 Oct 17. PMID 12410472
- [Background] Patel R. Clinical impact of vancomycin-resistant enterococci. J Antimicrob Chemother. 2003 Jun;51 Suppl 3:iii13-21. doi: 10.1093/jac/dkg272. PMID 12801938
- [Background] Kreman T, Hu J, Pottinger J, Herwaldt LA. Survey of long-term-care facilities in Iowa for policies and practices regarding residents with methicillin-resistant Staphylococcus aureus or vancomycin-resistant enterococci. Infect Control Hosp Epidemiol. 2005 Oct;26(10):811-5. doi: 10.1086/502498. PMID 16276955
- [Background] Bryce EA, Tiffin SM, Isaac-Renton JL, Wright CJ. Evidence of delays in transferring patients with methicillin-resistant Staphylococcus aureus or vancomycin-resistant Enterococcus to long-term-care facilities. Infect Control Hosp Epidemiol. 2000 Apr;21(4):270-1. doi: 10.1086/501757. PMID 10782590
- [Background] Baden LR, Thiemke W, Skolnik A, Chambers R, Strymish J, Gold HS, Moellering RC Jr, Eliopoulos GM. Prolonged colonization with vancomycin-resistant Enterococcus faecium in long-term care patients and the significance of "clearance". Clin Infect Dis. 2001 Nov 15;33(10):1654-60. doi: 10.1086/323762. Epub 2001 Oct 10. PMID 11595985
- [Background] Dunne C. Adaptation of bacteria to the intestinal niche: probiotics and gut disorder. Inflamm Bowel Dis. 2001 May;7(2):136-45. doi: 10.1097/00054725-200105000-00010. PMID 11383587
- [Background] Vanderhoof JA, Young RJ. Current and potential uses of probiotics. Ann Allergy Asthma Immunol. 2004 Nov;93(5 Suppl 3):S33-7. doi: 10.1016/s1081-1206(10)61730-9. PMID 15562872
- [Background] McFarland LV. Meta-analysis of probiotics for the prevention of antibiotic associated diarrhea and the treatment of Clostridium difficile disease. Am J Gastroenterol. 2006 Apr;101(4):812-22. doi: 10.1111/j.1572-0241.2006.00465.x. PMID 16635227
- [Background] Hickson M, D'Souza AL, Muthu N, Rogers TR, Want S, Rajkumar C, Bulpitt CJ. Use of probiotic Lactobacillus preparation to prevent diarrhoea associated with antibiotics: randomised double blind placebo controlled trial. BMJ. 2007 Jul 14;335(7610):80. doi: 10.1136/bmj.39231.599815.55. Epub 2007 Jun 29. PMID 17604300
- [Background] Manley KJ, Fraenkel MB, Mayall BC, Power DA. Probiotic treatment of vancomycin-resistant enterococci: a randomised controlled trial. Med J Aust. 2007 May 7;186(9):454-7. doi: 10.5694/j.1326-5377.2007.tb00995.x. PMID 17484706
- [Background] Hendrix CW, Hammond JM, Swoboda SM, Merz WG, Harrington SM, Perl TM, Dick JD, Borschel DM, Halczenko PW, Pelz RK, Rocco LE, Conway JE, Brower RG, Lipsett PA. Surveillance strategies and impact of vancomycin-resistant enterococcal colonization and infection in critically ill patients. Ann Surg. 2001 Feb;233(2):259-65. doi: 10.1097/00000658-200102000-00016. PMID 11176133
- [Background] Carmeli Y, Eliopoulos G, Mozaffari E, Samore M. Health and economic outcomes of vancomycin-resistant enterococci. Arch Intern Med. 2002 Oct 28;162(19):2223-8. doi: 10.1001/archinte.162.19.2223. PMID 12390066
- [Background] Patel R, Allen SL, Manahan JM, Wright AJ, Krom RA, Wiesner RH, Persing DH, Cockerill FR, Thompson RL. Natural history of vancomycin-resistant enterococcal colonization in liver and kidney transplant recipients. Liver Transpl. 2001 Jan;7(1):27-31. doi: 10.1053/jlts.2001.20784. PMID 11150418
- [Background] Montecalvo MA, de Lencastre H, Carraher M, Gedris C, Chung M, VanHorn K, Wormser GP. Natural history of colonization with vancomycin-resistant Enterococcus faecium. Infect Control Hosp Epidemiol. 1995 Dec;16(12):680-5. doi: 10.1086/647041. PMID 8683085
- [Background] Roghmann MC, Qaiyumi S, Schwalbe R, Morris JG Jr. Natural history of colonization with vancomycin-resistant Enterococcus faecium. Infect Control Hosp Epidemiol. 1997 Oct;18(10):679-80. doi: 10.1086/647510. No abstract available. PMID 9350457
- [Background] Borriello SP, Hammes WP, Holzapfel W, Marteau P, Schrezenmeir J, Vaara M, Valtonen V. Safety of probiotics that contain lactobacilli or bifidobacteria. Clin Infect Dis. 2003 Mar 15;36(6):775-80. doi: 10.1086/368080. Epub 2003 Mar 5. PMID 12627362
- [Background] Gorbach SL. Probiotics and gastrointestinal health. Am J Gastroenterol. 2000 Jan;95(1 Suppl):S2-4. doi: 10.1016/s0002-9270(99)00806-0. PMID 10634218
- [Background] Vanderhoof JA. Probiotics: future directions. Am J Clin Nutr. 2001 Jun;73(6):1152S-1155S. doi: 10.1093/ajcn/73.6.1152S. PMID 11393194
- [Background] Vanderhoof JA, Whitney DB, Antonson DL, Hanner TL, Lupo JV, Young RJ. Lactobacillus GG in the prevention of antibiotic-associated diarrhea in children. J Pediatr. 1999 Nov;135(5):564-8. doi: 10.1016/s0022-3476(99)70053-3. PMID 10547243
- [Background] Alvarez-Olmos MI, Oberhelman RA. Probiotic agents and infectious diseases: a modern perspective on a traditional therapy. Clin Infect Dis. 2001 Jun 1;32(11):1567-76. doi: 10.1086/320518. Epub 2001 May 4. PMID 11340528
- [Background] Sartor RB. Probiotic therapy of intestinal inflammation and infections. Curr Opin Gastroenterol. 2005 Jan;21(1):44-50. PMID 15687884
- [Background] Saxelin M, Chuang NH, Chassy B, Rautelin H, Makela PH, Salminen S, Gorbach SL. Lactobacilli and bacteremia in southern Finland, 1989-1992. Clin Infect Dis. 1996 Mar;22(3):564-6. doi: 10.1093/clinids/22.3.564. PMID 8852980
- [Background] Rayes N, Seehofer D, Theruvath T, Schiller RA, Langrehr JM, Jonas S, Bengmark S, Neuhaus P. Supply of pre- and probiotics reduces bacterial infection rates after liver transplantation--a randomized, double-blind trial. Am J Transplant. 2005 Jan;5(1):125-30. doi: 10.1111/j.1600-6143.2004.00649.x. PMID 15636620
- [Background] Rayes N, Seehofer D, Hansen S, Boucsein K, Muller AR, Serke S, Bengmark S, Neuhaus P. Early enteral supply of lactobacillus and fiber versus selective bowel decontamination: a controlled trial in liver transplant recipients. Transplantation. 2002 Jul 15;74(1):123-7. doi: 10.1097/00007890-200207150-00021. PMID 12134110
- [Background] Osterlund P, Ruotsalainen T, Korpela R, Saxelin M, Ollus A, Valta P, Kouri M, Elomaa I, Joensuu H. Lactobacillus supplementation for diarrhoea related to chemotherapy of colorectal cancer: a randomised study. Br J Cancer. 2007 Oct 22;97(8):1028-34. doi: 10.1038/sj.bjc.6603990. Epub 2007 Sep 25. PMID 17895895
- [Background] Delia P, Sansotta G, Donato V, Messina G, Frosina P, Pergolizzi S, De Renzis C, Famularo G. Prevention of radiation-induced diarrhea with the use of VSL#3, a new high-potency probiotic preparation. Am J Gastroenterol. 2002 Aug;97(8):2150-2. doi: 10.1111/j.1572-0241.2002.05946.x. No abstract available. PMID 12190202
- [Background] Rautio M, Jousimies-Somer H, Kauma H, Pietarinen I, Saxelin M, Tynkkynen S, Koskela M. Liver abscess due to a Lactobacillus rhamnosus strain indistinguishable from L. rhamnosus strain GG. Clin Infect Dis. 1999 May;28(5):1159-60. doi: 10.1086/514766. No abstract available. PMID 10452653
- [Background] Mackay AD, Taylor MB, Kibbler CC, Hamilton-Miller JM. Lactobacillus endocarditis caused by a probiotic organism. Clin Microbiol Infect. 1999 May;5(5):290-292. doi: 10.1111/j.1469-0691.1999.tb00144.x. No abstract available. PMID 11856270
- [Background] Land MH, Rouster-Stevens K, Woods CR, Cannon ML, Cnota J, Shetty AK. Lactobacillus sepsis associated with probiotic therapy. Pediatrics. 2005 Jan;115(1):178-81. doi: 10.1542/peds.2004-2137. PMID 15629999
- [Background] Kunz AN, Noel JM, Fairchok MP. Two cases of Lactobacillus bacteremia during probiotic treatment of short gut syndrome. J Pediatr Gastroenterol Nutr. 2004 Apr;38(4):457-8. doi: 10.1097/00005176-200404000-00017. No abstract available. PMID 15085028
- [Background] De Groote MA, Frank DN, Dowell E, Glode MP, Pace NR. Lactobacillus rhamnosus GG bacteremia associated with probiotic use in a child with short gut syndrome. Pediatr Infect Dis J. 2005 Mar;24(3):278-80. doi: 10.1097/01.inf.0000154588.79356.e6. PMID 15750472
- [Background] Klare I, Konstabel C, Werner G, Huys G, Vankerckhoven V, Kahlmeter G, Hildebrandt B, Muller-Bertling S, Witte W, Goossens H. Antimicrobial susceptibilities of Lactobacillus, Pediococcus and Lactococcus human isolates and cultures intended for probiotic or nutritional use. J Antimicrob Chemother. 2007 May;59(5):900-12. doi: 10.1093/jac/dkm035. Epub 2007 Mar 16. PMID 17369278